CLINICAL TRIAL: NCT00494260
Title: Intergenerational Transmission of Illness Behavior
Brief Title: Managing Recurrent Abdominal Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HD036069-07 (NIH)
Record Dates: First submitted 2007-06-28; First posted 2007-06-29 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Abdominal Pain
Keywords: recurrent abdominal pain; illness behavior; social learning; cognitive behavioral therapy
MeSH Terms: conditions — Abdominal Pain; Illness Behavior | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Social learning and cognitive behavioral therapy (SLCBT) (Experimental): The SLCBT condition consists of 3 main components: 1.) relaxation training, 2.) working with parent and child to modify family responses to illness and wellness behaviors, and 3.) cognitive restructuring to address and alter dysfunctional cognitions regarding symptoms and their implications for functioning through cognitive therapy techniques.
  Interventions: Behavioral: Social Learning and Cognitive Behavioral Therapy (SLCBT)
- Education Support (ES) (Active Comparator): The ES condition focuses on education about GI system anatomy and function, information about the United States Department of Agriculture nutrition guidelines, and additional food-related information such as how to read food product labels. The ES condition was developed to provide a credible alternative condition that would control for therapist and patient time and attention.
  Interventions: Behavioral: Education Support (ES)

INTERVENTIONS:
Behavioral: Social Learning and Cognitive Behavioral Therapy (SLCBT) — The SLCBT condition consists of 3 main components: 1.) relaxation training, 2.) working with parent and child to modify family responses to illness and wellness behaviors, and 3.) cognitive restructuring to address and alter dysfunctional cognitions regarding symptoms and their implications for functioning through cognitive therapy techniques
  Arms: Social learning and cognitive behavioral therapy (SLCBT)
Behavioral: Education Support (ES) — The ES condition focuses on education about GI system anatomy and function, information about the United States Department of Agriculture nutrition guidelines, and additional food-related information such as how to read food product labels. The ES condition was developed to provide a credible alternative condition that would control for therapist and patient time and attention.
  Arms: Education Support (ES)

SUMMARY:
The purpose of this study is to evaluate the efficacy of a social learning and cognitive behavior therapy approach for treating children with Recurrent Abdominal Pain (RAP).

DETAILED DESCRIPTION:
Recurrent Abdominal Pain (RAP) is one of many disorders in adults and children for which there is no identifiable organic or physiological cause, yet which is associated with illness behavior that has significant societal and personal costs. Although 10-15% of children have RAP, there is at present no accepted medical or behavioral treatment for it. We have conducted a series of studies that suggests that illness behavior is, at least in part, learned during childhood when parents model sick role behavior or respond to their children's somatic complaints in a way that encourages or reinforces sick role behavior. The goal of this project is to evaluate the efficacy of a social learning and cognitive behavior therapy approach for treating children with RAP.

The study is a randomized clinical trial. Children with RAP are assigned to one of two treatment conditions: 1) a social learning and cognitive behavior therapy condition (SLCBT) or 2) an education and support condition (ES). The SLCBT protocol teaches parents and children cognitive-behavioral methods such as relaxation and coping for managing RAP pain and stress. Patients and parents in the ES condition receive educational information regarding nutrition and the gastrointestinal system. Both treatment arms consist of three sessions with a mental health professional, each one week apart.

Study families are recruited from physicians in the community and through community flyers and newsletters. Outcome measures are collected at baseline, end of treatment, and at follow-up evaluations conducted three, six and 12 months later. Measures are designed to assess: RAP symptoms, health care utilization, psychological symptoms, school absences, functional disabilities, and family stress).

Primary Hypothesis: Children in the SLCBT condition will exhibit a greater decrease in symptoms of RAP and related maladaptive behaviors and cognitions than children in a comparison condition.

ELIGIBILITY:
Inclusion Criteria:

* child experienced at least 3 episodes of abdominal pain over a 3-month period which affected his/her activities
* primary caregiver willing and able to complete questionnaires
* child aged 7-17
* child has lived with the primary caregiver full-time for at least the past 5 years and for at least half of his/her lifetime

Exclusion Criteria:

* positive physical or laboratory findings which would explain the child's abdominal pain
* chronic disease
* major surgery in past year
* developmental disabilities that require full-time special education or impair ability to respond
* inability to comprehend English

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2003-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
symptoms of recurrent abdominal pain | measured one week following treatment and again in 3, 6 and 12 months
disability | measured one week following treatment and again in 3, 6 and 12 months

SECONDARY OUTCOMES:
parent behaviors | measured one week following treatment and again in 3, 6 and 12 months
child coping behaviors | measured one week following treatment and again in 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rona Levy, PhD, Principal Investigator — School of Social Work, University of Washington
Locations (2):
- United States (2):
  - Goryeb Children's Hospital/ Atlantic Health System, Morristown, New Jersey
  - University of Washington/ Children's Hospital and Regional Medical Center, Seattle, Washington

REFERENCES:
- [Background] Levy RL, Whitehead WE, Walker LS, Von Korff M, Feld AD, Garner M, Christie D. Increased somatic complaints and health-care utilization in children: effects of parent IBS status and parent response to gastrointestinal symptoms. Am J Gastroenterol. 2004 Dec;99(12):2442-51. doi: 10.1111/j.1572-0241.2004.40478.x. PMID 15571594
- [Background] Levy RL, Whitehead WE, Von Korff MR, Feld AD. Intergenerational transmission of gastrointestinal illness behavior. Am J Gastroenterol. 2000 Feb;95(2):451-6. doi: 10.1111/j.1572-0241.2000.01766.x. PMID 10685749
- [Derived] Levy RL, Langer SL, Walker LS, Romano JM, Christie DL, Youssef N, DuPen MM, Ballard SA, Labus J, Welsh E, Feld LD, Whitehead WE. Twelve-month follow-up of cognitive behavioral therapy for children with functional abdominal pain. JAMA Pediatr. 2013 Feb;167(2):178-84. doi: 10.1001/2013.jamapediatrics.282. PMID 23277304